CLINICAL TRIAL: NCT07151313
Title: Efficacy of Bee Venom Phonophoresis in Treating Chronic Sinusitis: A Double-Blind Randomized Controlled Trial
Brief Title: Efficacy of Bee Venom Phonophoresis in Treating Chronic Sinusitis:
Acronym: BEE-SONIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, lecturer, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU.REC.2025(48H)
Record Dates: First submitted 2025-08-10; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Chronic Sinusitis; Acute Sinusitis; Rhinosinusitis
Keywords: Sinusitis; Rhinosinusitis, Chronic; Rhinosinusitis, Acute
MeSH Terms: conditions — Rhinosinusitis; Sinusitis; Bronchiolitis Obliterans Syndrome | interventions — Standard of Care; Nasal Decongestants

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Double Blind (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bee Venom Phonophoresis (Experimental): Participants receive bee venom phonophoresis therapy three times per week for the study duration. Ultrasound parameters set at 1 MHz frequency, low-to-moderate intensity, applied in circular or linear motion for 5-10 minutes per sinus. Bee venom is mixed with ultrasound coupling gel and applied to targeted sinus areas.
  Intervention Name: Bee Venom Phonophoresis
  Interventions: Device: Bee Venom Phonophoresis; Biological: Bee Venom Phonophoresis
- Standard Care (Placebo Comparator): Participants receive standard medical treatment for sinusitis, consisting of oral decongestants and saline nasal irrigation, according to local clinical guidelines.
  Interventions: Drug: Standard Care (oral decongestants + saline nasal irrigation)

INTERVENTIONS:
Device: Bee Venom Phonophoresis — Ultrasound therapy device
  Arms: Bee Venom Phonophoresis
Drug: Standard Care (oral decongestants + saline nasal irrigation) — (oral decongestants + saline nasal irrigation)
  Arms: Standard Care
Biological: Bee Venom Phonophoresis — bee venom extract prepared for topical use)
  Arms: Bee Venom Phonophoresis

SUMMARY:
This double-blind, randomized controlled trial (BEE-SONIC) aims to evaluate the efficacy of bee venom phonophoresis in the treatment of chronic sinusitis. Thirty adult patients (aged 18-65 years) with clinically diagnosed chronic or acute sinusitis will be randomized into two groups: the intervention group will receive bee venom phonophoresis using low-to-moderate intensity ultrasound, while the control group will receive standard care consisting of oral decongestants and saline nasal irrigation. Primary outcomes include improvement in symptom severity (SNOT-22, Visual Analog Scale) and quality of life (SF-33). Secondary outcomes include reduction in facial pain, nasal congestion, and patient satisfaction. Data will be collected at baseline, midpoint, and post-intervention, and analyzed using paired t-tests and ANOVA. The study has received ethics approval from Sinai University's Human Research Ethics Committee, and informed consent will be obtained from all participants.

DETAILED DESCRIPTION:
Chronic sinusitis is a prevalent condition characterized by persistent inflammation of the paranasal sinuses, often resulting in nasal congestion, facial pain, and reduced quality of life. Conventional treatments, including antibiotics, nasal corticosteroids, and decongestants, may provide limited relief and can be associated with adverse effects. Bee venom possesses anti-inflammatory and analgesic properties, while phonophoresis - the use of ultrasound to enhance transdermal drug delivery - can facilitate deeper tissue penetration of therapeutic agents. Combining bee venom with phonophoresis may represent a novel, non-invasive treatment strategy for chronic sinusitis.

This randomized, double-blind, controlled clinical trial (BEE-SONIC) will enroll 30 adult participants aged 18-65 years with clinically diagnosed chronic or acute sinusitis. Participants will be randomly assigned to one of two groups: the intervention group will receive bee venom phonophoresis three times per week for the study duration, and the control group will receive standard care comprising oral decongestants and saline nasal irrigation. Ultrasound parameters for the intervention will be set at a frequency of 1 MHz and low-to-moderate intensity, with each sinus treated for 5-10 minutes per session.

The primary outcome measures are changes in symptom severity assessed by the Sino-Nasal Outcome Test (SNOT-22) and Visual Analog Scale (VAS) for pain, as well as quality of life measured by the SF-33 questionnaire. Secondary outcomes include reductions in facial pain and nasal congestion, and patient satisfaction with the treatment. Data will be collected at baseline, mid-intervention, and post-intervention. Statistical analysis will include descriptive statistics, paired t-tests, and ANOVA, with a significance threshold set at p < 0.05.

Ethics approval has been obtained from Sinai University's Human Research Ethics Committee, and all participants will provide written informed consent prior to study enrollment. Confidentiality will be maintained throughout the trial, and findings will be disseminated through peer-reviewed publications and conference presentations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Clinical diagnosis of chronic sinusitis (symptoms ≥ 12 weeks) or acute sinusitis confirmed by an otolaryngologist.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Known allergy or hypersensitivity to bee venom or bee products.
* Skin conditions (e.g., eczema, dermatitis, open wounds) over the area of ultrasound application.
* Severe comorbid medical conditions (e.g., uncontrolled asthma, autoimmune disease, malignancy).
* Pregnancy or breastfeeding.
* Use of systemic corticosteroids, antibiotics, or other medications that may significantly alter sinusitis symptoms within 4 weeks prior to enrollment.
* Participation in another clinical trial within the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in Sinusitis Symptom Severity | Baseline (day 0), mid-intervention (week 2), and end of intervention (week 4).
  Measured using the Sino-Nasal Outcome Test (SNOT-22) questionnaire, which assesses nasal, facial, and functional symptoms on a 0-5 Likert scale (total score range: 0-110; higher scores indicate worse symptoms).
Change in Pain Intensity | Baseline (day 0), mid-intervention (week 2), and end of intervention (week 4).
  Measured using a Visual Analog Scale (VAS) for facial pain, ranging from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline (day 0), mid-intervention (week 2), and end of intervention (week 4).
  Measured using the SF-36 questionnaire, which assesses physical, emotional, and social health domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai university, Cairo, Egypt